CLINICAL TRIAL: NCT06706414
Title: Novel Treatment of Some Men With Non-Obstructive Azoospermia (NT-NOA): A Clinical Interventional Study
Brief Title: NT-NOA - Novel Treatment of Some Men With Non-Obstructive Azoospermia
Acronym: NT-NOA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, Head of Research Department Endocrinology, Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-512996-11-00; 2024-512996-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Denosumab; Letrozole; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Denosumab (Experimental): Subcutaneous injection with 60 mg Denosumab once
  Interventions: Drug: Denosumab (Prolia); Drug: Letrozole (Aromatase Inhibitors)

INTERVENTIONS:
Drug: Denosumab (Prolia) — Subcutaneous injection with 60 mg Denosumab once
Drug: Letrozole (Aromatase Inhibitors) — Letrozole oral tablet 2.5 mg once daily

SUMMARY:
This clinical interventional study aims to assess whether treatment with denosumab in combination with letrozole can improve sperm production in infertile men with non-obstructive azoospermia selected by serum anti-mullerian hormone (AMH) as a positive predictive biomarker.

DETAILED DESCRIPTION:
Infertility is a health issue worldwide with more than 15% of couples experiencing infertility. Male factors contribute in 50% of all cases and is the sole cause in 30% of all infertile couples . Treatment options for the male infertility are limited and only specific conditions like varicocele and hypogonadotropic hypogonadism can be effectively treated with surgery and hormonal stimulation, respectively. However, for the remaining 90% of infertile men, no treatment options exist. Instead, their female partners must undergo fertility treatment.

Men with the most pronounced impairment of semen quality, men with azoospermia, have no sperm in the ejaculate and are classically divided into obstructive azoospermia (OA) and non-obstructive azoospermia (NOA), with the ladder being the most common. These men needs to have surgery performed for sperm retrieval with either testicular sperm aspiration (TESA), testicular sperm extraction (TESE) or micro testicular sperm extraction (microTESE) in order to have a chance of becoming biological fathers. The chance of successful sperm retrieval in men with OA is close to 100%, whereas men with NOA have a significantly lower chance with only around 10-40% being successful. This is due to the vast difference in etiology between men with OA and NOA. Even with a successful surgical intervention only half of the cases will result in a live birth, leaving the majority of men with NOA no chance of becoming biological fathers. Therefore, novel treatment options for even a minor sub-group of these men are warranted.

RANKL is a ligand for the receptor activator of nuclear factor kappa beta (RANK), and their pathway plays a prominent role in the regulation of bone metabolism. The binding of RANKL to RANK on osteoclast precursors induces osteoclast maturation and activation, thereby stimulating bone resorption, and regulates cell cycle i.e., proliferation, differentiation, and apoptosis. Osteoprotegerin (OPG) is a secreted decoy receptor that controls RANKL-RANK interaction by binding RANKL and inhibits activation of RANK and preventing osteoclast differentiation and activation.

Denosumab, a drug used in millions of patients worldwide under trade names Prolia® and Xgeva®, inhibits the RANKL pathway and is used to treat osteoporosis and bone metastases. The drug's mechanism of action inhibits RANKL and thus inhibits bone resorption through reduced osteoclast activation. This reduces the loss of bone mineral density (BMD), which reduces the risk of bone loss and thereby the risk of fracture and osteoporosis. Denosumab has been shown in several clinical studies to be a safe and effective drug in both women and men and has been in clinical use in both sexes for many years. As Denosumab has a teratogenic effect, pharmacokinetic studies in both monkeys and healthy men were performed before approval of the drug as a treatment for osteoporosis in men. These studies showed that Denosumab concentration in semen does not pose a risk to the fetus during sexual intercourse with the pregnant woman and therefore is safe to use for the suggested infertility indication as there is no risk of fetal transmission.

The investigators have also shown that RANKL also influences germ cell apoptosis, differentiation, and proliferation in mice and humans. This indicates that the RANKL system could be a potential direct regulator of spermatogenesis, and thus highlighting that the drug Denosumab, a RANKL inhibitor, commonly used to treat osteoporosis, may be used for medical treatment of men with decreased sperm production. The effects of denosumab in vitro were supported by a pilot intervention study in 12 infertile men, which showed that denosumab either had a highly beneficial or detrimental effect on sperm production. This implies that only a sub-group of infertile men should be offered this treatment and these men should be identified by, preferably, a simple and accessible biomarker.

Therefore, the investigators are currently conducting two randomized clinical trials "First In Treating Infertility (FITMI)" and "Novel Approach for Oligospermia (NAPO) to explore whether denosumab can improve semen quality in infertile men selected by serum AMH, but already have sperm concentration between 2 mio/mL - 20 mio/mL (FITMI) and 0.01 mio/mL - 2 mio/mL (NAPO). These are both important studies, but still leaves out men with no sperm in the ejaculate, azoospermic patients. Therefore, there is a need for a trial adressing these patients for a potential novel treatment option.

NT-NOA is a single-center, sponsor-investigator-initiated, interventional trial, Following successful completion of screening procedures, subjects will all receive denosumab 60 mg s.c. and Letrozole oral tablet 2.5 mg once daily. Participants will all initiate letrozole treatment 14 days prior to the denosumab injection and will continue until the TESE procedure. The study will be carried out at the Division of Translational Endocrinology, Copenhagen University Hospital, Herlev, Copenhagen, Denmark.

The investigators believe it is of clinical relevance to treat 10 patients with denosumab in combination with letrozole for 1 of them to achieve sperm production, however, it is difficult to estimate. Ideally 50% of the treated participants will have sperm suitable for ART post intervention. By including 16 patients, there will be sufficient power to determine if combination therapy with denosumab and letrozole induces a clinically relevant effect on spermatogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Infertile men ≥ 18 years and < 60 years of age with azoospermia with normal semen volume (> 0.9 mL) verified by minimum 2 semen samples.
* No identifiable cause of obstruction.
* Testis size (Prader Orchidometer) ≤ 15 mL on both sides in patients where no prior TESE is available
* Serum AMH levels ≥5 pmol/L.

Exclusion Criteria:

* Chronic diseases, defined as diagnosis where signs, symptoms, and treatment imply an expected long duration and lack of a cure, such as diabetes mellitus, metabolism disorders, osteoporosis, colitis, etc.
* Chromosome anomalies e.g. Klinefelter Syndrome, XX male
* AZFa/b/c microdeletions besides b2/b3 og gr/gr
* Detected CFTR mutation
* Men with current or previous malignancies, or at potential risk of testicular cancer after baseline examination and ultrasound will be excluded
* Men with hypocalcemia at baseline, defined as albumin corrected calcium < 2.17 mmol/L or total calcium < 2.14 mmol/L
* Serum vitamin D (25OHD) levels < 25 nmol/L
* estimated Glomerular Filtration Rate (eGFR) < 60 mL/min/1,73 m2
* Insufficient dental status
* Hypersensitivity to latex, Denosumab, or to any of the excipients (acetic acid, sodium hydroxide, Sorbitol (E420), Polysorbate 20) will be excluded.
* Serum Inhibin B < 5 pg/mL
* Androgen replacement therapy
* Hypogonadotropic hypogonadism
* BMI ≥ 35 kg/m2

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Sperm in the semen sample or TESE on day 90 | Day 80 (semen sample) and 90 (TESE) after inclusion
  Finding of sperm in the semen sample (day 80) or TESE (day 90), that subsequently will be compared with prior TESE if available.

SECONDARY OUTCOMES:
The change in expression of proliferation (KI-67, PCNA) and apoptosis (cPARP, TUNEL assay) markers in TESE tissue at day 90 compared to prior TESE if available | Day 90 after inclusion
  TESE
The number of participants with sperm in the ejaculate (sperm pr. milliliter) assessed by semen samples delivered on day 14 | Day 14 after inclusion
  Semen sample
The number of participants with sperm in the ejaculate (sperm pr. milliliter) assessed by semen samples delivered on day 80 | Day 80 after inclusion
  Semen sample
The number of pregnancies achieved by sperm from the ejaculate or by TESE | Day 180 after inclusion
  Survey
The change in serum levels of reproductive hormones (FSH, LH, AMH, Inhibin B og INSL3) on day 14 | Day 14 after inclusion
  Serum sample
The change in serum levels of reproductive hormones (FSH, LH, AMH, Inhibin B og INSL3) on day 80 | Day 80 after inclusion
  Serum sample
The change in serum levels of sex steroids (Testosterone, Estradiol and SHBG) on day 14 | Day 14 after inclusion
  Serum sample
The change in serum levels of sex steroids (Testosterone, Estradiol and SHBG) on day 80 | Day 80 after inclusion
  Serum sample
The change in seminal fluid levels of reproductive hormones (AMH, Inhibin B, INSL3) on day 14 | Day 14 after inclusion
  Seminal fluid
The change in seminal fluid levels of reproductive hormones (AMH, Inhibin B, INSL3) on day 80 | Day 80 after inclusion
  Seminal fluid
The change in the endocrine gonadal function (Inhibin B/FSH ratio, Testosterone/LH ratio and AMH/testosterone ratio) on day 14 | Day 14 after inclusion
  Serum sample
The change in the endocrine gonadal function (Inhibin B/FSH ratio, Testosterone/LH ratio and AMH/testosterone ratio) on day 80 | Day 80 after inclusion
  Serum sample

OTHER OUTCOMES:
The change in seminal fluid levels of RANKL, OPG, AMH and Inhibin B on day 14 | Day 14 after inclusion
  Seminal fluid
The change in seminal fluid levels of RANKL, OPG, AMH and Inhibin B on day 80 | Day 80 after inclusion
  Seminal fluid
The change in serum levels of minerals (calcium, phosphate, magnesium, zink, bikarbonate, citrate) on day 14 | Day 14 after inclusion
  Serum
The change in serum levels of minerals (calcium, phosphate, magnesium, zink, bikarbonate, citrate) on day 80 | Day 80 after inclusion
  Serum
The change in seminal fluid levels of minerals (calcium, phosphate, magnesium, zink, bikarbonate, citrate) on day 14 | Day 14 after inclusion
  Seminal fluid
The change in seminal fluid levels of minerals (calcium, phosphate, magnesium, zink, bikarbonate, citrate) on day 80 | Day 80 after inclusion
  Seminal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Christian F.S. Jensen, MD, PhD., Principal Investigator — Department of Urology, Herlev and Gentofte Hospital
Locations (1):
- Division of Translational Endocrinology, Department of Endocrinology and Internal Medicine, Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huynh AL, Baker ST, Stewardson AJ, Johnson DF. Denosumab-associated hypocalcaemia: incidence, severity and patient characteristics in a tertiary hospital setting. Pharmacoepidemiol Drug Saf. 2016 Nov;25(11):1274-1278. doi: 10.1002/pds.4045. Epub 2016 Jun 3. PMID 27255807
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Main KM. Testicular dysgenesis syndrome: an increasingly common developmental disorder with environmental aspects. Hum Reprod. 2001 May;16(5):972-8. doi: 10.1093/humrep/16.5.972. PMID 11331648
- [Background] Toulis KA, Anastasilakis AD. Increased risk of serious infections in women with osteopenia or osteoporosis treated with denosumab. Osteoporos Int. 2010 Nov;21(11):1963-4. doi: 10.1007/s00198-009-1145-1. Epub 2009 Dec 15. No abstract available. PMID 20012939
- [Background] Anastasilakis AD, Toulis KA, Goulis DG, Polyzos SA, Delaroudis S, Giomisi A, Terpos E. Efficacy and safety of denosumab in postmenopausal women with osteopenia or osteoporosis: a systematic review and a meta-analysis. Horm Metab Res. 2009 Oct;41(10):721-9. doi: 10.1055/s-0029-1224109. Epub 2009 Jun 17. PMID 19536731
- [Background] Bone HG, Chapurlat R, Brandi ML, Brown JP, Czerwinski E, Krieg MA, Mellstrom D, Radominski SC, Reginster JY, Resch H, Ivorra JA, Roux C, Vittinghoff E, Daizadeh NS, Wang A, Bradley MN, Franchimont N, Geller ML, Wagman RB, Cummings SR, Papapoulos S. The effect of three or six years of denosumab exposure in women with postmenopausal osteoporosis: results from the FREEDOM extension. J Clin Endocrinol Metab. 2013 Nov;98(11):4483-92. doi: 10.1210/jc.2013-1597. Epub 2013 Aug 26. PMID 23979955
- [Background] Lamy O, Stoll D, Aubry-Rozier B, Rodriguez EG. Stopping Denosumab. Curr Osteoporos Rep. 2019 Feb;17(1):8-15. doi: 10.1007/s11914-019-00502-4. PMID 30659428
- [Background] Uebelhart B, Rizzoli R, Ferrari SL. Retrospective evaluation of serum CTX levels after denosumab discontinuation in patients with or without prior exposure to bisphosphonates. Osteoporos Int. 2017 Sep;28(9):2701-2705. doi: 10.1007/s00198-017-4080-6. Epub 2017 May 24. PMID 28540505
- [Background] Bekker PJ, Holloway DL, Rasmussen AS, Murphy R, Martin SW, Leese PT, Holmes GB, Dunstan CR, DePaoli AM. A single-dose placebo-controlled study of AMG 162, a fully human monoclonal antibody to RANKL, in postmenopausal women. J Bone Miner Res. 2004 Jul;19(7):1059-66. doi: 10.1359/JBMR.040305. Epub 2004 Mar 1. PMID 15176987
- [Background] Blomberg Jensen M, Andreassen CH, Jorgensen A, Nielsen JE, Juel Mortensen L, Boisen IM, Schwarz P, Toppari J, Baron R, Lanske B, Juul A. RANKL regulates male reproductive function. Nat Commun. 2021 Apr 23;12(1):2450. doi: 10.1038/s41467-021-22734-8. PMID 33893301
- [Background] Bussiere JL, Pyrah I, Boyce R, Branstetter D, Loomis M, Andrews-Cleavenger D, Farman C, Elliott G, Chellman G. Reproductive toxicity of denosumab in cynomolgus monkeys. Reprod Toxicol. 2013 Dec;42:27-40. doi: 10.1016/j.reprotox.2013.07.018. Epub 2013 Jul 22. PMID 23886817
- [Background] Sohn W, Lee E, Kankam MK, Egbuna O, Moffat G, Bussiere J, Padhi D, Ng E, Kumar S, Slatter JG. An open-label study in healthy men to evaluate the risk of seminal fluid transmission of denosumab to pregnant partners. Br J Clin Pharmacol. 2016 Feb;81(2):362-9. doi: 10.1111/bcp.12798. Epub 2015 Dec 5. PMID 26447647
- [Background] Boonen S, Adachi JD, Man Z, Cummings SR, Lippuner K, Torring O, Gallagher JC, Farrerons J, Wang A, Franchimont N, San Martin J, Grauer A, McClung M. Treatment with denosumab reduces the incidence of new vertebral and hip fractures in postmenopausal women at high risk. J Clin Endocrinol Metab. 2011 Jun;96(6):1727-36. doi: 10.1210/jc.2010-2784. Epub 2011 Mar 16. PMID 21411557
- [Background] Papapoulos S, Chapurlat R, Libanati C, Brandi ML, Brown JP, Czerwinski E, Krieg MA, Man Z, Mellstrom D, Radominski SC, Reginster JY, Resch H, Roman Ivorra JA, Roux C, Vittinghoff E, Austin M, Daizadeh N, Bradley MN, Grauer A, Cummings SR, Bone HG. Five years of denosumab exposure in women with postmenopausal osteoporosis: results from the first two years of the FREEDOM extension. J Bone Miner Res. 2012 Mar;27(3):694-701. doi: 10.1002/jbmr.1479. PMID 22113951
- [Background] Polyzos SA, Singhellakis PN, Naot D, Adamidou F, Malandrinou FC, Anastasilakis AD, Polymerou V, Kita M. Denosumab treatment for juvenile Paget's disease: results from two adult patients with osteoprotegerin deficiency ("Balkan" mutation in the TNFRSF11B gene). J Clin Endocrinol Metab. 2014 Mar;99(3):703-7. doi: 10.1210/jc.2013-3762. Epub 2014 Jan 16. PMID 24433001
- [Background] Schwarz P, Rasmussen AQ, Kvist TM, Andersen UB, Jorgensen NR. Paget's disease of the bone after treatment with Denosumab: a case report. Bone. 2012 May;50(5):1023-5. doi: 10.1016/j.bone.2012.01.020. PMID 22586699
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Terpos E. RANKL inhibition for the management of patients with benign metabolic bone disorders. Expert Opin Investig Drugs. 2009 Aug;18(8):1085-102. doi: 10.1517/13543780903048929. PMID 19558335
- [Background] Makras P, Polyzos SA, Papatheodorou A, Kokkoris P, Chatzifotiadis D, Anastasilakis AD. Parathyroid hormone changes following denosumab treatment in postmenopausal osteoporosis. Clin Endocrinol (Oxf). 2013 Oct;79(4):499-503. doi: 10.1111/cen.12188. Epub 2013 Apr 1. PMID 23452098
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Anastasilakis CD, Makras P. Long-term treatment of osteoporosis: safety and efficacy appraisal of denosumab. Ther Clin Risk Manag. 2012;8:295-306. doi: 10.2147/TCRM.S24239. Epub 2012 Jun 19. PMID 22767993
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Kwiecinski GG, Petrie GI, DeLuca HF. Vitamin D is necessary for reproductive functions of the male rat. J Nutr. 1989 May;119(5):741-4. doi: 10.1093/jn/119.5.741. PMID 2723823
- [Background] Uhland AM, Kwiecinski GG, DeLuca HF. Normalization of serum calcium restores fertility in vitamin D-deficient male rats. J Nutr. 1992 Jun;122(6):1338-44. doi: 10.1093/jn/122.6.1338. PMID 1588451
- [Background] Blomberg Jensen M. Vitamin D and male reproduction. Nat Rev Endocrinol. 2014 Mar;10(3):175-86. doi: 10.1038/nrendo.2013.262. Epub 2014 Jan 14. PMID 24419359